CLINICAL TRIAL: NCT02355821
Title: Comparative Effects of Moxonidine and Bisoprolol on Bone Metabolism, Vascular and Cellular Markers of Aging, Blood Pressure in Hypertensive Postmenopausal Women (COMPASS)
Brief Title: Comparative Effects of Moxonidine on Bone Metabolism, Vascular and Cellular Aging in Hypertensive Postmenopausal Women
Acronym: COMPASS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Research Center for Preventive Medicine (Other Government)
Responsible Party: Sponsor
Organization: National Medical Research Center for Therapy and Preventive Medicine (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: MOXOC001
Record Dates: First submitted 2015-01-13; First posted 2015-02-04 (Estimated); Results first posted 2021-09-01 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Osteopenia; Arterial Hypertension
Keywords: cellular aging; vascular aging; bone metabolism; collagen type 1 C-telopeptide; nuclear factor kappa-B ligand (RANKL); pulse wave velocity; telomerase activity
MeSH Terms: conditions — Bone Diseases, Metabolic; Hypertension; Osteopetrosis, mild autosomal recessive form | interventions — moxonidine; Bisoprolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Moxonidine (Experimental): 0.4 mg moxonidine QD titration up to 0.6 mg moxonidine BID
  Interventions: Drug: Moxonidine
- Bisoprolol (Active Comparator): 5 mg Bisoprolol QD titration up to 7.5 mg Bisoprolol BID
  Interventions: Drug: Bisoprolol

INTERVENTIONS:
Drug: Moxonidine — 0.4 mg moxonidine QD titration up to 0.6 mg moxonidine BID Other Names:perindopril 10 mg/day (optional); losartan 50 mg/day (optional); calcium carbonate; vitamin D
  Other Names: Physiotens
  Arms: Moxonidine
Drug: Bisoprolol — 5 mg Bisoprolol QD titration up to 7.5 mg Bisoprolol BID Other Names: perindopril 10 mg/day (optional); losartan 50 mg/day (optional); calcium carbonate; vitamin D
  Arms: Bisoprolol

SUMMARY:
This study evaluates the effect of moxonidine versus bisoprolol on collagen type 1 C-telopeptide in postmenopausal female patients with arterial hypertension and osteopenia.

DETAILED DESCRIPTION:
Several experimental studies have demonstrated that moxonidine may lower the activity of Na+- independent Cl-/bicarbonate exchanger (anion exchanger, AE) which plays an essential role in viability of osteoclasts that are crucial for bone resorption. The suppression of AE proteins activity has been proven to inhibit osteoclast activity and reduce bone resorption whereas the moxonidine molecule is known to reduce the AE protein activity. Therefore, the results of experimental studies have shown the ability of moxonidine to inhibit bone resorption through its effect on the osteoclast activity.

Published data contain information on positive effects of beta-blockers on the bone tissue condition. There are data which clearly demonstrate a positive effect of beta-blockers on bone mass.

The proposed trial is a comprehensive study of moxonidine effects on processes of cellular and vascular aging as well as bone metabolism.

ELIGIBILITY:
Inclusion Criteria:

1. Female with age 45 years and older.
2. Postmenopausal (absence of menstrual periods for a minimum of 12 months) at the moment of Informed Consent sign.
3. Arterial hypertension grade I / II per ESH/ESC 2013 guidelines (diastolic pressure ≥ 90 and <110 mm Hg, systolic pressure ≥140 and <180 mm Hg).
4. Not achieving BP targets <140/90 mmHg either during antihypertensive therapy or naive.
5. Absence of moxonidine or bisoprolol treatment at least 6 months before the study
6. Osteopenia of lumbar spine and/or proximal part of the femur (osteoporosis T-score from -1 to -2.5 standard deviations [SD]) by X-Ray densitometry.
7. Signed Informed Consent for participation in the study

   -

Exclusion Criteria:

1. Hypersensitivity to moxonidine, bisoprolol or any other ingredient of the respective formulations
2. Any Contraindications for moxonidine, bisoprolol
3. Osteoporosis (Т-score below - 2.5 SD).
4. Primary or secondary hyperparathyroidism.
5. Paget's disease of bones.
6. History of low traumatic bone fractures.
7. Malabsorption syndrome.
8. History of gastro-intestinal surgery.
9. Severe disturbance of peripheral circulation.
10. Raynaud's disease.
11. Symptomatic (secondary) hypertension (caused by any primary internal diseases)
12. Morbid obesity (BMI over 40 kg/m2).
13. Symptoms of estrogen deficiency such as hot flushes, nights sweat, vaginal dryness
14. Administration of any hormone-replacement therapy (HRT) or intake of isoflavones
15. Secondary hypogonadism.
16. Sistolic BP ≥180 mm Hg and/or Diastolic BP ≥110 mm Hg.
17. Clinical presentations of cardiovascular disease: coronary heart disease (CHD), history of stroke, transient ischemic attack (TIA), Charcot's syndrome.
18. Severe heart failure.
19. Hemodynamically significant congenital heart disease.
20. Heart rhythm disorders which require permanent use of any antiarrhythmic medications (including β-adrenoblockers and calcium antagonists).
21. Diabetes mellitus of any genesis.
22. Severe liver failure.
23. Severe kidney failure including patients on dialysis
24. Thyroid diseases accompanied by functional disorders (thyrotoxicosis or uncompensated hypothyroidism).
25. Alcohol and drug abuse.
26. Patients with oncological diseases diagnosed within 5 years before IC execution.
27. Inability of the patient to comprehend the essence of the program and to provide his/her consent for participation in the program.
28. Patients with any condition, which in the opinion of the Investigator makes the patient unsuitable for inclusion based on clinical judgment.
29. Corticosteroid therapy
30. Participation in any other clinical study during the whole course of this investigation including participation in a study within 30 days prior to providing the informed consent for this trial

    -

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2015-04; Primary Completion 2018-06-15 (Actual); Study Completion 2018-07-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Olga N Tkacheva, Professor, Principal Investigator — tkacheva@rambler.ru
Locations (1):
- National Research Center for Preventive Medicine, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Moxonidine | Bisoprolol
Started | 57 | 57
Completed | 57 | 57
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Moxonidine | Bisoprolol | Total
Number analyzed (Participants) | 57 | 57 | 114
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 32 | 32 | 64
  >=65 years | 25 | 25 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.96 (9.1) | 60.5 (9.1) | 62 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 57 | 114
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 57 | 57 | 114
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Russia | 57 | 57 | 114
Bone resorption marker (collagen type 1 C-telopeptide) [Median (Inter-Quartile Range); unit: ng/ml] | 0.4 [0.3 to 0.5] | 0.4 [0.3 to 0.6] | 0.4 [0.3 to 0.6]

OUTCOME MEASURES:

1. Primary Outcome: Collagen Type 1 C-telopeptide
Description: Changes in Median (Inter-Quartile Range) of the bone resorption marker (collagen type 1 C-telopeptide) at the end of the study from the baseline are evaluated in comparison between the groups
Time Frame: baseline (Visit 1) and 12 months (Visit 4)
Measure: Median (Inter-Quartile Range); unit: ng/ml
Arm/Group | Moxonidine | Bisoprolol
Number analyzed (Participants) | 57 | 57
ng/ml
  Baseline | 0.4 [0.3 to 0.5] | 0.4 [0.3 to 0.6]
  12 months | 0.3 [0.2 to 0.4] | 0.4 [0.3 to 0.5]

2. Secondary Outcome: Osteocalcin
Description: Changes in Median (Inter-Quartile Range) values of the bone synthesis marker (osteocalcin) at the end of the study (V4) from the baseline (V1) and to compare the values between the groups.
Time Frame: baseline (Visit 1) and 12 months (Visit 4)
Measure: Median (Inter-Quartile Range); unit: ng/ml
Arm/Group | Moxonidine | Bisoprolol
Number analyzed (Participants) | 57 | 57
ng/ml
  Baseline | 18.2 [12.4 to 21.9] | 19.4 [12.4 to 26.2]
  12 months | 19.6 [15.4 to 23.5] | 18.7 [12.8 to 22.79]

3. Secondary Outcome: Receptor Activator of Nuclear Factor Kappa-B Ligand (RANKL).
Description: Changes in Median (Inter-Quartile Range) values of the receptor activator of nuclear factor kappa-B ligand (RANKL) at final visit versus baseline level in comparison between the groups
Time Frame: baseline (Visit 1) and 12 months (Visit 4)
Measure: Median (Inter-Quartile Range); unit: pmol/ml
Arm/Group | Moxonidine | Bisoprolol
Number analyzed (Participants) | 57 | 57
pmol/ml
  Baseline | 0.109 [0.06 to 0.18] | 0.133 [0.06 to 0.182]
  12 month | 0.09 [0.05 to 0.17] | 0.111 [0.07 to 0.163]

4. Secondary Outcome: Bone Mineral Density (BMD) Using Control Dual-energy X-ray Absorptiometry
Description: Changes in Median (Inter-Quartile Range) values of Bone mineral density (BMD) at final visit versus baseline level using control dual-energy X-ray absorptiometry and in comparison between the groups
Time Frame: 12 months
Population: Total hip BMD
Measure: Median (Inter-Quartile Range); unit: g/cm2
Arm/Group | Moxonidine | Bisoprolol
Number analyzed (Participants) | 57 | 57
g/cm2
  Baseline | -1.0 [-1.7 to -0.2] | -0.55 [-1.3 to -0.2]
  12 months | -0.6 [-0.9 to -0.1] | -1.2 [-1.9 to -0.75]

5. Secondary Outcome: Telomerase Activity
Description: Changes in Median (Inter-Quartile Range) telomerase activity at final visit versus baseline level in comparison between the groups Telomerase activity is measured in arbitrary units. Currently, there are no established reference values for telomerase activity in the world. Its activity is considered high or low in relation to the median.
Time Frame: baseline (Visit 1) and 12 months (Visit 4)
Measure: Median (Inter-Quartile Range); unit: arbitrary units
Arm/Group | Moxonidine | Bisoprolol
Number analyzed (Participants) | 57 | 57
arbitrary units
  Baseline | 0.87 [0.16 to 1.18] | 0.89 [0.16 to 1.15]
  12 months | 1.15 [0.74 to 1.59] | 0.64 [0.46 to 1.01]

6. Secondary Outcome: Pulse Wave Velocity (PWV)
Description: Changes in mean pulse wave velocity (PWV) at final visit versus baseline level and in comparison between the groups
Time Frame: baseline (Visit 1) and 12 months (Visit 4)
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | Moxonidine | Bisoprolol
Number analyzed (Participants) | 57 | 57
m/s
  Baseline | 10.35 (2.56) | 10.36 (2.47)
  12 months | 10.05 (2.29) | 11.26 (2.6)

7. Secondary Outcome: Intima-media Thickness (IMT)
Description: Changes in mean intima-media thickness (IMT) at final visit in comparison between the groups.
Time Frame: baseline (Visit 1) and 12 months (Visit 4)
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Moxonidine | Bisoprolol
Number analyzed (Participants) | 57 | 57
mm
  Baseline | 0.98 (0.17) | 0.98 (0.15)
  12 months | 0.77 (0.14) | 0.88 (0.16)

8. Secondary Outcome: THe Number (Percentage) of the Treatment Responders
Description: Proportion of the treatment responders (defined as the proportion (%) of patients who achieved target blood pressure <140/90 mmHg) after 8 and 48 weeks of the investigated treatment (V2, V3 and V4) and to compare the values between the groups.
Time Frame: baseline (Visit 1) and 12 months (Visit 4)
Measure: Count of Participants; unit: Participants
Arm/Group | Moxonidine | Bisoprolol
Number analyzed (Participants) | 57 | 57
Participants | 55 | 53

9. Secondary Outcome: Number of Participants With Adverse Events (AE)
Description: Number of Participants with Adverse Events (AE)
Time Frame: baseline (Visit 1) and 12 months (Visit 4)
Measure: Count of Participants; unit: Participants
Arm/Group | Moxonidine | Bisoprolol
Number analyzed (Participants) | 57 | 57
Participants | 3 | 3

ADVERSE EVENTS:
Time Frame: baseline (Visit 1) and 12 months (Visit 4)
Arm/Group | Moxonidine | Bisoprolol
All-Cause Mortality (participants affected / at risk) | 0/57 | 0/57
Serious Adverse Events (participants affected / at risk) | 0/57 | 0/57
Other Adverse Events (participants affected / at risk) | 3/57 | 3/57
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Moxonidine (N=57) | Bisoprolol (N=57)
headache (General disorders) | 2 (2) | 1 (1) — headache
cough (General disorders) | 0 (0) | 2 (2)
Dry mouth (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2014-12-12): https://cdn.clinicaltrials.gov/large-docs/21/NCT02355821/Prot_SAP_ICF_000.pdf